CLINICAL TRIAL: NCT04598477
Title: An Open-Label, Multicenter, Follow-up Trial of ARGX-113-1904 to Evaluate the Safety, Tolerability, and Efficacy of Efgartigimod PH20 SC in Patients With Pemphigus
Brief Title: A Study to Assess the Long-term Safety and Efficacy of a Subcutaneous Formulation of Efgartigimod PH20 SC in Adults With Pemphigus (Vulgaris or Foliaceus)
Acronym: ADDRESS+
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on the lack of observed efficacy in the primary study ARGX-113-1904, the sponsor decided to discontinue the open-label extension study.
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-1905
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pemphigus Vulgaris; Pemphigus Foliaceus
MeSH Terms: conditions — Pemphigus | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- efgartigimod PH20 SC (Experimental): patients receiving efgartigimod PH20 SC on top of prednisone
  Interventions: Biological: efgartigimod PH20 SC; Drug: prednisone

INTERVENTIONS:
Biological: efgartigimod PH20 SC — Subcutaneous injection of efgartigimod using rHuPH20 (PH20) as a permeation enhancer
Drug: prednisone — Oral prednisone tablets

SUMMARY:
This was a prospective, multicenter, open label extension (OLE) trial on the efficacy, safety, patient outcome measures, tolerability, immunogenicity, PK and PD of efgartigimod PH20 SC in adult PV or PF participants, who participated in antecedent trial ARGX-113-1904. This trial provided extension of efgartigimod PH20 SC treatment and retreatment options for participants who had been randomized to efgartigimod PH20 SC treatment arm in the trial ARGX-113-1904, and first treatment of efgartigimod PH20 SC and retreatment options for participants who had been randomized to the placebo arm in trial ARGX-113-1904. The participants could also receive concomitant prednisone therapy. Investigators could increase or decrease the prednisone dose based on protocol-specified criteria.

Trial ARGX-113-1905 evaluated the ability to (further) taper prednisone therapy and achieve Clinical Remission (CR) off therapy (CRoff), the ability to achieve CR and CR on minimal therapy (CRmin) for participants who had not yet achieved CR or CRmin, and the ability to treat flare; it also assessed patient outcome measures and the safety, PD, PK and immunogenicity of efgartigimod PH20 SC over the duration of trial.

Study duration: Up to 60 weeks for participants who receive IMP administration up to 52 weeks and with a follow-up period of 8 weeks after the last IMP administration

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the requirements of the trial, to provide written informed consent (including consent for the use and disclosure of research-related health information), willingness and ability to comply with the trial protocol procedures (including required trial visits).
2. The participant participated in trial ARGX-113-1904 and completed the study or has the defined criteria for rollover.
3. Contraceptive use by men and women should be consistent with local regulations regarding the methods for contraception for those participating in clinical trials and:

   1. Male participants:

      Male participants must agree to use an acceptable method of contraception as described in the protocol, from signing the ICF until the last dose of the study drug.
   2. Female participants

Women of childbearing potential (WOCBP) must:

* have a negative urine pregnancy test at baseline before the IMP can be administered,
* agree to use a highly effective or acceptable contraception method (as described in the protocol), which should be maintained at minimum until after the last dose of IMP

Exclusion Criteria:

1. Pregnant and lactating women and those intending to become pregnant during the trial.
2. Participants with clinical evidence of other significant serious disease or participants who recently underwent or have planned a major surgery during the period of the trial, or any other condition in the opinion of the investigator, that could confound the results of the trial or put the participant at undue risk.
3. Known hypersensitivity to any of the components of the administered treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (127):
- United States (17):
  - Investigator site 115 - US0010086, Birmingham, Alabama
  - Investigator site 89 - US0010091, Scottsdale, Arizona
  - Investigator site 124 - US0010092, Redwood City, California
  - Investigator site 1 - US0010087, Boca Raton, Florida
  - Investigator site 90 - US0010117, Miami, Florida
  - Investigator site 91 - US0010109, Orlando, Florida
  - Investigator site 126 - US0010090, Minneapolis, Minnesota
  - Investigator site 111 - US0010098, St Louis, Missouri
  - Investigator site 10 - US0010088, Buffalo, New York
  - Investigator site 76 - US0010096, Durham, North Carolina
  - Investigator site 30 - US0010094, Cleveland, Ohio
  - Investigator site 84 - US0010089, Philadelphia, Pennsylvania
  - Investigator site 103 - US0010097, Philadelphia, Pennsylvania
  - Investigator site 125 - US0010107, Dallas, Texas
  - Investigator site 87 - US0010084, Dripping Springs, Texas
  - Investigator site 88 - US0010114, Houston, Texas
  - Investigator site 44 - US0010106, Norfolk, Virginia
- Australia (3):
  - Investigator site 15 - AU0610006, Sydney, New South Wales
  - Investigator site 11 - AU0610007, Parkville, Victoria
  - Investigator site 92 - AU0610013, Melbourne
- Bulgaria (5):
  - Investigator site 17 - BG3590012, Pleven
  - Investigator site 18 - BG3590013, Plovdiv
  - Investigator site 2 - BG3590010, Sofia
  - Investigator site 16 - BG3590009, Sofia
  - Investigator site 3 - BG3590011, Sofia
- China (13):
  - Investigator site 101 - CN0860017, Beijing
  - Investigator site 107 - CN0860018, Chengdu
  - Investigator site 118 - CH0860027, Chongqing
  - Investigator site 120 - CH0860023, Fuzhou
  - Investigator site 119 - CH0860022, Guangzhou
  - Investigator site 116 - CH0860053, Guangzhou
  - Investigator site 100 - CN0860021, Guanzhou
  - Investigator site 113 - CN0860024, Nanjing
  - Investigator site 102 - CN0860020, Shanghai
  - Investigator site 99 - CN0860016, Shanghai
  - Investigator site 112 - CN0860019, Wuhan
  - Investigator site 121 - CH0860025, Wuhan
  - Investigator site 117 - CH0860026, Zhengzhou
- France (4):
  - Investigator site 77 - FR0330028, Bobigny
  - Investigator site 60 - FR0330027, La Tronche
  - Investigator site 108 - FR0330029, Rouen
  - Investigator site 51 - FR0330026, Saint-Etienne
- Georgia (4):
  - Investigator site 78 - GE9950014, Tbilisi
  - Investigator site 127 - GE9950030, Tbilisi
  - Investigator site 32 - GE9950013, Tbilisi
  - Investigator site 31 - GE9950015, Tbilisi
- Germany (10):
  - Investigator site 45 - DE0490029, Berlin
  - Investigator site 34 - DE0490030, Dresden
  - Investigator site 33 - DE0490024, Frankfurt am Main
  - Investigator site 53 - DE0490023, Freiburg im Breisgau
  - Investigator site 35 - DE0490028, Kiel
  - Investigator site 20 - DE0490002, Lübeck
  - Investigator site 52 - DE0490001, Marburg
  - Investigator site 19 - DE0490025, Tübingen
  - Investigator site 93 - DE0490027, Ulm
  - Investigator site 4 - DE0490026, Würzburg
- Greece (6):
  - Investigator site 21 - GR030004, Athens
  - Investigator site 37 - GR030006, Athens
  - Investigator site 54 - GR0300001, Athens
  - Investigator site 22 - GR030003, Chaïdári
  - Investigator site 36 - GR0300002, Thessaloniki
  - Investigator site 23 - GR030005, Thessaloniki
- Hungary (3):
  - Investigator site 6 - HU0360003, Debrecen
  - Investigator site 5 - HU0360001, Pécs
  - Investigator site 24 - HU0360002, Szeged
- India (4):
  - Investigator site 65 - IN0910002, Ahmedabad
  - Investigator site 94 - IN0910001, Chandigarh
  - Investigator site 79 - IN0910004, Lucknow
  - Investigator site 80 - IN0910003, Nagpur
- Investigator site 85 - IL9720002, Tel Aviv, Israel
- Italy (7):
  - Investigator site 95 - IT0390039, Catania
  - Investigator site 38 - IT0390031, Florence
  - Investigator site 81 - IT0390030, Genova
  - Investigator site 55 - IT0390038, Perugia
  - Investigator site 12 - IT0390006, Roma
  - Investigator site 25 - IT-0390005, Roma
  - Investigator site 61 - IT0390040, Siena
- Japan (10):
  - Investigator site 82 - JP0810046, Aichi
  - Investigator site 68 - JP0810040, Hiroshima
  - Investigator site 66 - JP0810042, Kofu
  - Investigator site 69 - JP0810050, Kurume
  - Investigator site 73 - JP0810047, Okayama
  - Investigator site 70 - JP0810041, Okayama
  - Investigator site 71 - JP0810049, Osaka
  - Investigator site 72 - JP0810045, Sapporo
  - Investigator site 114 - JP0810067, Sendai
  - Investigator site 67 - JP0810043, Tokyo
- Poland (5):
  - Investigator site 27 - PL0480027, Katowice
  - Investigator site 56 - PL0480032, Lodz
  - Investigator site 86 - PL0480036, Poznan
  - Investigator site 28 - PL0480025, Rzeszów
  - Investigator site 26 - PL0480028, Wroclaw
- Romania (3):
  - Investigator site 97 - RO0400013, Bucharest
  - Investigator 96 - RO0400014, Cluj-Napoca
  - Investigator site 98 - RO0400015, Iași
- Russia (8):
  - Investigator site 40 - RU0070035, Chelyabinsk
  - Investigator site 48 - RU0070029, Kazan'
  - Investigator site 49 - RU0070030, Krasnodar
  - Investigator site 39 - RU0070032, Rostov-on-Don
  - Investigator site 46 - RU0070031, Saint Petersburg
  - Investigator site 50 - RU0070034, Saint Petersburg
  - Investigator site 47 - RU0070028, Saratov
  - Investigator site 41 - RU0070033, Yekaterinburg
- Serbia (4):
  - Investigator site 109 - RS3810011, Belgrade
  - Investigator site 110 - RS3810010, Belgrade
  - Investigator site 105 - RS3810012, Niš
  - Investigator site 104 - RS3810009, Novi Sad
- Spain (8):
  - Investigator site 62 - ES0340026, Barcelona
  - Investigator site 13 - ES0340032, Barcelona
  - Investigator site 122 - ES0340053, Granada
  - Investigator site 59 - ES0340034, Madrid
  - Investigator site 42 - ES0340025, Madrid
  - Investigator site 7 - ES0340029, Madrid
  - Investigator site 57 - ES0340027, Madrid
  - Investigator site 58 - ES0340028, Seville
- Turkey (Türkiye) (3):
  - Investigator site 64 - TR0900020, Gaziantep
  - Investigator site 63 - TR0900012, Istanbul
  - Investigator site 74 - TR0900011, Istanbul
- Ukraine (6):
  - Investigator site 75 - UA3800017, Dnipro
  - Investigator site 29 - UA3800023, Ivano-Frankivsk
  - Investigator site 14 - UA3800020, Kyiv
  - Investigator site 8 - UA3800019, Kyiv
  - Investigator site 43 - UA3800021, Lviv
  - Investigator site 9 - UA3800018, Zaporizhzhia
- United Kingdom (3):
  - Investigator site 106 - UK0440021, Birmingham
  - Investigator site 83 - UK0440022, Bristol
  - Investigator site 123 - UK0440037, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated early based on the lack of observed efficacy in antecedent ARGX-113-1904. A total of 183 participants rolled over from ARGX-113-1904. Of these, 57 participants had a CRmin status (complete remission on minimal prednisone therapy) at rollover of which 34 participants did not receive efgartigimod PH20 SC in this ARGX-113-1905 study.
Pre-assignment Details: Two main analysis sets were analyzed in the outcome measures: Roll-over set includes all participants regardless of whether they received efgartigimod PH20 SC treatment during this study. Safety set includes participants who received at least 1 dose of efgartigimod PH20 SC during this study.
  Additional restrictions to the analysis set might apply in the different outcome measures. These are described in the analysis population descriptions.
Groups:
- Efgartigimod-efgartigimod PH20 SC: Participants who received efgartigimod PH20 SC in antecedent study ARGX-113-1904.
- Placebo-efgartigimod PH20 SC: Participants who received placebo PH20 SC in antecedent study ARGX-113-1904.
Period: Overall Study
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Started | 123 | 60
Completed | 64 | 23
Not Completed | 59 | 37
Not completed — Adverse Event | 2 | 0
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 7 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Requires Prohibited Medication | 0 | 1
Not completed — Study Terminated by Sponsor | 18 | 12
Not completed — Withdrawal by Subject | 16 | 12
Not completed — Other | 15 | 8

BASELINE CHARACTERISTICS:
Population: Roll-over set
Groups:
- Total: Total of all reporting groups
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC | Total
Number analyzed (Participants) | 123 | 60 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.40) | 52.4 (13.02) | 50.8 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 32 | 93
  Male | 62 | 28 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 40 | 9 | 49
  Black or African American | 1 | 2 | 3
  White | 81 | 47 | 128
  Other | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 120 | 56 | 176

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (TEAE), Adverse Events of Special Interest (AESI), and Serious Adverse Events (SAE)
Description: Incidence rates were calculated as 100 × n/PYFU. PYFU=participant-years of follow-up. The safety data sets includes participants with pemphigus vulgaris (PV) and pemphigus foliaceus (PF).
Time Frame: Up to 60 weeks
Population: Safety set
Measure: Number; unit: number of events x 100/PYFU
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 101 | 48
number of events x 100/PYFU
  Treatment-Emergent Adverse Event (TEAE) | 116.4 | 113.0
  Adverse Event of Special Interest (AESI) | 72.0 | 69.3
  Serious Adverse Event (SAE) | 24.5 | 14.6

2. Secondary Outcome: Proportion of Participants With Pemphigus Vulgaris (PV) and Pemphigus Foliaceus (PF) Who Achieve CRmin
Description: CRmin defined as the absence of new lesions and complete healing of established lesions while the participant was receiving prednisone at ≤10 mg/day for at least 8 weeks.
Time Frame: Up to 60 weeks
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 101 | 48
Participants | 55 | 26

3. Secondary Outcome: Proportion of Participants With Pemphigus Vulgaris (PV) Who Achieve CRmin
Description: CRmin (complete clinical remission on minimal prednisone therapy) defined as the absence of new lesions and complete healing of established lesions while the participant was receiving prednisone at ≤10 mg/day for at least 8 weeks.
Time Frame: Up to 60 weeks
Population: Safety set - Participants with PV
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 86 | 41
Participants | 47 | 22

4. Secondary Outcome: Time to DC in Participants With PV and PF
Description: Disease Control (DC) defined as absence of new lesions and the start of healing of established lesions
Time Frame: Up to 52 weeks
Population: Safety set - Participants with status DC at the roll-over visit were not included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 26 | 17
days | 8.5 [8.0 to 15.0] | 15.0 [8.0 to 22.0]

5. Secondary Outcome: Time to CR in Participants With PV and PF
Description: CR (Complete clinical remission) defined as the absence of new lesions and complete healing of established lesions
Time Frame: Up to 52 weeks
Population: Safety set - Participants with status CR at the roll-over visit were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 61 | 34
Days | 66.0 [43.0 to 182.0] | 71.0 [41.0 to 100.0]

6. Secondary Outcome: Time to CRmin in Participants With PV and PF
Description: as for outcome 2
Time Frame: Up to 52 weeks
Population: Safety set - Participants with status CRmin at the roll-over visit were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 83 | 43
days | 229.0 [161.0 to NA] — The upper limit of 95% CI could not be reported because of insufficient number of participants with events. | 169.0 [141.0 to 322.0]

7. Secondary Outcome: Time to CRoff in Participants With PV and PF
Description: Complete remission off therapy (CRoff) is defined as the absence of new and established lesions completely healed while the patient is receiving no prednisone therapy for at least 8 weeks.
Time Frame: Up to 52 weeks
Population: Safety set - Participants with status CRoff at the roll-over visit were not included in this analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 83 | 43
days | NA [NA to NA] — The median survival time (95% CI) could not be calculated because the survival probability (95% CI) exceeded 50% at the longest time | NA [NA to NA] — The median survival time (95% CI) could not be calculated because the survival probability (95% CI) exceeded 50% at the longest time

8. Secondary Outcome: Time to Flare After CRmin in Participants With PV and PF
Description: CRmin defined as defined as the absence of new lesions and complete healing of established lesions while the participant was receiving prednisone at ≤10 mg/day for at least 8 weeks.
Time Frame: Up to 52 weeks
Population: Safety set - Only participants who achieved CRmin were considered for the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 42 | 23
days | 339.0 [223.0 to NA] — The upper limit of the 95% CI could not be reported because of insufficient number of participants with events. | 168.0 [64.0 to NA] — The upper limit of 95% CI could not be reported because of insufficient number of participants with events.

9. Secondary Outcome: Rate of Treatment Failure in Participants With PV and PF
Description: The absence of DC with oral prednisone 1.5 mg/kg/day for a minimum of 3 weeks, or absence of DC due to prednisone-related SAE, or flare before CRmin resulting in withdrawal of the participant.
Time Frame: Up to 52 weeks
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 101 | 48
Participants | 3 | 1

10. Secondary Outcome: Number of Flares in Participants With PV and PF
Description: A flare is defined as the appearance of 3 or more new lesions in a 4-week period that do not heal spontaneously within 1 week or the extension, of established lesions in a participant who had achieved DC.
Time Frame: Up to 60 weeks
Population: Roll-over set - Only participants who achieved DC were considered for the analysis.
Measure: Mean (Standard Deviation); unit: Flares
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 122 | 59
Flares | 0.8 (1.03) | 0.7 (0.79)

11. Secondary Outcome: Normalized Cumulative Prednisone Dose in Participants With PV and PF
Description: Normalized Cumulative prednisone dose (NCPD, mg/kg/day) is the average daily intake of all weight-adjusted prednisone doses received during the study, taking into account the number of days in study
Time Frame: Up to 60 weeks
Population: Roll-over set - For participants that do not achieve CRmin (or CRoff), NCPD until CRmin (or CRoff) is not calculated
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
Number analyzed (Participants) | 123 | 60
mg/kg/day | 0.212 (0.2018) | 0.241 (0.2401)

ADVERSE EVENTS:
Time Frame: Up to 60 weeks
Description: Participants who rolled over from the antecedent study ARGX-113-1904, and received at least 1 dose of efgartigimod PH20 SC during this ARGX-113-1905 study (Safety set). Laboratory abnormalities were reported as AEs.
Arm/Group | Efgartigimod-efgartigimod PH20 SC | Placebo-efgartigimod PH20 SC
All-Cause Mortality (participants affected / at risk) | 0/101 | 1/48
Serious Adverse Events (participants affected / at risk) | 16/101 | 4/48
Other Adverse Events (participants affected / at risk) | 46/101 | 19/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod-efgartigimod PH20 SC (N=101) | Placebo-efgartigimod PH20 SC (N=48)
ANAL FISTULA (Gastrointestinal disorders) | 1 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 2 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
REFLUX GASTRITIS (Gastrointestinal disorders) | 1 | 0
DISEASE PROGRESSION (General disorders) | 2 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
EPIGLOTTITIS (Infections and infestations) | 1 | 0
LUNG ABSCESS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 0
SKIN INFECTION (Infections and infestations) | 0 | 1
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
WOUND (Injury, poisoning and procedural complications) | 1 | 0
BLOOD IMMUNOGLOBULIN G DECREASED (Investigations) | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PEMPHIGUS (Skin and subcutaneous tissue disorders) | 3 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 1 | 0
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod-efgartigimod PH20 SC (N=101) | Placebo-efgartigimod PH20 SC (N=48)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 | 3
TACHYCARDIA (Cardiac disorders) | 1 | 3
INJECTION SITE ERYTHEMA (General disorders) | 4 | 3
COVID-19 (Infections and infestations) | 12 | 5
FOLLICULITIS (Infections and infestations) | 5 | 1
NASOPHARYNGITIS (Infections and infestations) | 5 | 1
ORAL CANDIDIASIS (Infections and infestations) | 6 | 0
URINARY TRACT INFECTION (Infections and infestations) | 5 | 2
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 7 | 1
BLOOD URIC ACID INCREASED (Investigations) | 5 | 0
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 6 | 0
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 5 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 5 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 2 | 3
HEADACHE (Nervous system disorders) | 3 | 4
HAEMATURIA (Renal and urinary disorders) | 2 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
Study was terminated prematurely by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT04598477/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT04598477/SAP_001.pdf